CLINICAL TRIAL: NCT03839225
Title: Effectiveness of a Community - Based Cross-sector Network for the Management of Mental Health Problems and Disorders Associated With Forced Displacement Due to Armed Conflict in the Municipality of Soacha - Cundinamarca
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad Nacional de Colombia (Other)
Collaborators: The University of Bath in England (Unknown); Sociedad Colombiana de Anestesiología y Reanimación (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: Soacha 1
Record Dates: First submitted 2018-11-22; First posted 2019-02-15 (Actual); Last update posted 2021-04-29 (Actual); Status verified 2021-04

CONDITIONS: Mental Disorder; Mental Disorder in Adolescence; Mental Problems; Mental Disorder in Infancy
MeSH Terms: conditions — Mental Disorders

STUDY DESIGN:
Intervention Model Description: A mixed study of before and after using quantitative and qualitative research techniques
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Children, Adolescents and Adults (Other): children, adolescents and adults who have been victims of the armed conflict in the municipalities of Soacha-Cundimanarca (Colombia)
  Interventions: Other: Community intervention

INTERVENTIONS:
Other: Community intervention — Community intervention will be built depending on contextual factors and will contain the following elements:
  * Cross-sector intervention, including sectors to define the intervention as "primary health care services, education services" (language, knowledge to prevent health problems and resilience strategies), family welfare units, "Integral Care and Reparation Unit for Victims" (UARIV), Ministry of Labour, national and international social support network, among others.
  * The leader will be chosen by the community, with the capabilities to coordinate the community-based network.
  * Mental health providers at the local level, who must develop psychosocial and mental diagnoses and interventions, based on experience and evidence, respectively. This team will include psychiatry, psychologists (one an expert in clinical psychology) and a community team involved in the implementation of mental interventions.

SUMMARY:
It is of great importance to generate interventions that help ensure greater inclusion and social participation of the population that was and is a victim of the armed conflict, especially in the post-conflict transition in Colombia, and to influence development in the post-accord period through relationships between groups and society. Therefore, the question for this investigation is, what is the effectiveness of a community-based cross-sector network for the management of mental problems and disorders associated with forced displacement due to armed conflict in the commune of Soacha - Cundinamarca, in order to contribute to inclusion and social participation in the post-accord period?

Objective: To design a community-based cross-sector network for the management of mental problems and disorders associated with forced displacement due to armed conflict in the commune of Soacha - Cundinamarca, in order to contribute to inclusion and social participation in the post-accord period in Colombia.

ELIGIBILITY:
Inclusion Criteria:

• Children (7 to 11 years old), adolescents (12 to 18 years old) and adults (>18 years old) who have been victims of the armed conflict in the municipalities of Soacha - Cundinamarca, occurring during the last 5 years prior to the start of the project

Exclusion Criteria:

• People with neurocognitive disorders

Ages: 7 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 299 (Actual)
Dates: Start 2018-11-01 (Actual); Primary Completion 2019-09-01 (Actual); Study Completion 2020-07-01 (Actual)

PRIMARY OUTCOMES:
Change from the measure of mental disorders, including depression, anxiety-related disorders, and somatoform disorders: adolescents and adults at 1 year (after Community - Based Cross-sector Network implementation) | Before (baseline) and 1 year after Community - Based Cross-sector Network implementation
  Scale: the Self-Reporting Questionnaire (SRQ) which were used in the 2015 National Mental Health Survey in Colombia. SRQ consists of 20 items indicative of non-psychotic mental disorders, each of the 20 items is scored 0 or 1. A score of 1 indicates that the symptom was present during the past month, a score of o indicates that the symptom was absent.
Change from the measure of Child mental health problems (between the ages of 5 and 15) at 1 year (after Community - Based Cross-sector Network implementation) | Before (baseline) and 1 year after Community - Based Cross-sector Network implementation
  Scale: Reporting Questionnaire for Children (RQC) is a 10-item instrument administered verbally to the caregivers of children. It has been shown to identify moderate to severe mental retardation, significant degrees of emotional or behavioral disorder, which adversely affect schooling or socialization, and psychotic disorders among children.
  The instrument is scored by placing an X in any of the two response options and is scored in a simple manner, assigning one (1) point for each positive response. The presence of only an affirmative answer is indicative of the presence of a mental health problem.
  A single positive item was considered an appropriate cut-off for screening cases and perhaps for pointing towards a particular disorder. The RQC has 88% sensitivity in identifying cases diagnosed by a psychiatrist using a diagnostic interview according to the DSM-IV
Change from depression measure (adolescents and adults) at 1 year (after Community - Based Cross-sector Network implementation) | Before (baseline) and 1 year after Community - Based Cross-sector Network implementation
  Scale: The PHQ-9 is the depression module, which scores each of the nine DSM-IV criteria as "0" (not at all) to "3" (nearly every day).
Change from Posttraumatic Stress Disorder (children, adolescents and adults) at 1 year (after Community - Based Cross-sector Network implementation) | Before (baseline) and 1 year after Community - Based Cross-sector Network implementation
  The POSTTRAUMATIC STRESS DISORDER CHECKLIST (PCL-5) is a 20-item self-report measure that assesses the 20 DSM-5 symptoms of PTSD. The PCL-5 has a variety of purposes, including Monitoring symptom change during and after treatment, Screening individuals for PTSD, and Making a provisional PTSD diagnosis.
  A total symptom severity score (range - 0-80) can be obtained by summing the scores for each of the 20 items. A PCL-5 cut-point score is 33. The test is designed in such a way that if an item is answered, it is scored "0" and the next question is followed. Now, if he answers affirmatively, the questions that follow the item are formulated to know the frequency. Sometimes scored with "1" and sometimes with "2", the total score is 60, a fact that reflects the frequency of the symptoms

SECONDARY OUTCOMES:
Change from the personal factors of resilience (adolescents and adults) at 1 year (after Community - Based Cross-sector Network implementation) | Before (baseline) and 1 year after Community - Based Cross-sector Network implementation
  Personal factors of resilience Scale (FPR-1) was developed to analyze the personal factors of resilience in a group of 113 women displaced by violence in Colombia.
  377/5000 It is a Likert scale, with three response options: in disagreement (1), neither agree nor disagree (2) and agree (3). Scores between 1 and 1.5 are considered a low level; scores between 1.6 and 2 are considered medium-low; scores between 2.1 and 2.5 medium-high; Scores between 2.6 and 3 indicate a high level for global resilience or for the specific dimension.
Change from the measure of the problem or risky substance use in Children, adolescents, and adults at 1 year (after Community - Based Cross-sector Network implementation) | Before (baseline) and 1 year after Community - Based Cross-sector Network implementation
  Scale: Alcohol, Smoking and Substance Involvement Screening Test (ASSIST) was developed for the World Health Organization (WHO) by an international group of substance abuse researchers to detect and manage substance use and related problems in primary and general medical care settings.
  A risk score is provided for each substance, and scores are grouped into low, moderate or high risk.
  Low risk: scores of 'three or less' ('10 or less' for alcohol) of presenting problems related to substance use Moderate risk: score between 4 and 26 '('11 and 26' for alcohol), although they may present some problems, they have a moderate risk of presenting health and other problems.
  High risk: score of '27 or more 'in any substance suggests that the user has a high risk of dependence on that substance and is probably having health, social, economic, legal and personal relationship problems as a result of the consumption of substances.
Change from the measure of Hazardous and harmful alcohol consumption (adolescents and adults) at 1 year (after Community - Based Cross-sector Network implementation) | Before (baseline) and 1 year after Community - Based Cross-sector Network implementation
  Scale: The Alcohol Use Disorders Identification Test (AUDIT) is a very reliable and simple screening tool which is sensitive to early detection of risky and high risk (or hazardous and harmful) drinking. It has three questions on alcohol consumption (1 to 3), three questions on drinking behaviour and dependence (4 to 6) and four questions on the consequences or problems related to drinking (7 to 10).
  Scores for each question range from 0 to 4, with the first response for each question (eg never) scoring 0, the second (eg less than monthly) scoring 1, the third (eg monthly) scoring 2, the fourth (eg weekly) scoring 3, and the last response (eg. daily or almost daily) scoring 4. For questions 9 and 10, which only have three responses, the scoring is 0, 2 and 4 (from left to right). A score of 8 or more is associated with harmful or hazardous drinking, a score of 13 or more in women, and 15 or more in men, is likely to indicate alcohol dependence.

OTHER OUTCOMES:
Change from the measure of Family Functioning at 1 year (after Community - Based Cross-sector Network implementation) | Before (baseline) and 1 year after Community - Based Cross-sector Network implementation
  The Family APGAR has frequently been utilized as a tool for assessing family function.
  The maximum score to obtain is 20/20 points; the score obtained by the family allows to classify it in 4 ranges of family functioning:
  * Good family functioning, with scores between 18 - 20
  * Mild family dysfunction, with scores between 14 - 17
  * Moderate family dysfunction with scores between 10 - 13
  * Severe family dysfunction with scores of 9 or less.
Change from the measure of Eating Attitudes (adolescents and adults) at 1 year (after Community - Based Cross-sector Network implementation) | Before (baseline) and 1 year after Community - Based Cross-sector Network implementation
  Eating Attitudes Test© (EAT-26) is a screening measure to help you determine whether you might have an eating disorder that needs professional attention. Scores greater than 20 indicate a need for further investigation by a qualified professional. Low scores (below 20) can still be consistent with serious eating problems, as a denial of symptoms can be a problem with eating disorders.
Change from the measure of Bullying (ages between 10 and 18 years) at 1 year (after Community - Based Cross-sector Network implementation) | Before (baseline) and 1 year after Community - Based Cross-sector Network implementation
  Scale to identify victims of bullying and measure the intensity of this way in students

CONTACTS AND LOCATIONS:
Locations (1):
- Facultad de Medicina, Universidad Nacional de Colombia, Bogotá, Colombia